CLINICAL TRIAL: NCT04145297
Title: A Phase I Trial of Ulixertinib (BVD-523) and Hydroxychloroquine in Patients with Advanced MAPK-Mutated Gastrointestinal Adenocarcinomas
Brief Title: Ulixertinib (BVD-523) and Hydroxychloroquine in Patients W Advanced MAPK-Mutated Gastrointestinal Adenocarcinomas
Acronym: UTAH
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: BioMed Valley Discoveries, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCI127114
Record Dates: First submitted 2019-10-28; First posted 2019-10-30 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Gastrointestinal Neoplasms
MeSH Terms: conditions — Gastrointestinal Neoplasms | interventions — ulixertinib; Hydroxychloroquine

STUDY DESIGN:
Intervention Model Description: Open-label dose escalation of Ulixertinib combined with fixed dose of hydroxychloroquine.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment: all patients (Experimental): Hydroxychloroquine will be provided as 200 mg tablets and will be self-administered by mouth twice daily.
  Ulixertinib will be provided as 150 mg capsules and will be self-administered twice daily by mouth at the assigned dose level. Both medications will be administered in 28-day cycles
  Interventions: Drug: Ulixertinib; Drug: Hydroxychloroquine

INTERVENTIONS:
Drug: Ulixertinib — Ulixertinib will be provided as 150 mg capsules and will be self-administered twice daily by mouth at the assigned dose level.
  Ulixertinib Dose Level 0 300 mg PO BID, Dose Level 1 (starting dose) 450 mg PO BID, Dose Level 2 600 mg PO BID,
  Medication will be administered in 28-day cycles
  Other Names: BVD-523
Drug: Hydroxychloroquine — Hydroxychloroquine will be provided as 200 mg tablets and will be self-administered by mouth twice daily. Fixed Dose 600mg POBID. Medication will be administered in 28-day cycles

SUMMARY:
Open-label dose escalation of Ulixertinib combined with fixed dose of hydroxychloroquine.

DETAILED DESCRIPTION:
This is an open-label Phase I basket trial designed to determine the phase 2 recommended dose of ulixertinib in combination hydroxychloroquine. The recommended phase 2 dose (RP2D) will be determined by using a standard 3+3 dose-escalation design with a minimum of 3 evaluable subjects accrued to dose level one and two. Should dose level one be deemed intolerable, enrollment will proceed at dose level 0. The RP2D will be affirmed according to the rules of the 3+3 dose-escalation scheme

ELIGIBILITY:
Inclusion Criteria:

* Male or female subject aged ≥ 18 years.
* Subject with histologically confirmed MAPK-mutated GI malignancies: KRAS, NRAS, HRAS, BRAFnon-V600, MEK, and ERK.
* Subject is willing to provide a baseline biopsy.
* Prior lines of therapy:

  * For patients with cholangiocarcinoma: subject must have progressed during or after one line of therapy.
  * For patients with pancreatic adenocarcinoma: the subject must have progressed during or after one line of therapy.
  * For patients with colorectal carcinoma: the subject must have progressed during or after two lines of therapy.
  * For patients with stomach or esophageal carcinoma: the subject must have progressed during or after two lines of therapy.
* Subject must have measurable disease by RECIST 1.1 criteria by CT or MRI.
* ECOG Performance Status ≤ 1.
* Adequate organ function as defined as:

  * Hematologic:

    * Absolute neutrophil count (ANC) ≥ 1500/mm3
    * Platelet count ≥ 100,000/mm3
    * Hemoglobin ≥ 10 g/dL
  * Hepatic:

    * Total Bilirubin ≤ 1.5x institutional upper limit of normal (ULN)
    * AST(SGOT)/ALT(SGPT) ≤ 3 × institutional ULN
    * Patients with liver metastases will be allowed to enroll with AST and ALT levels ≤ 5 x ULN.
  * Renal:

    * Estimated creatinine clearance ≥ 50 mL/min by Cockcroft-Gault formula:
    * Males: ((140-age)×weight[kg])/(serum creatinine [mg/dL]×72)
    * Females: (((140-age)×weight[kg])/(serum creatinine [mg/dL]×72))×0.85
* Evidence of post-menopausal status or negative urinary or serum pregnancy test for female pre-menopausal patients. Women will be considered post-menopausal if they have been amenorrheic for 12 months without an alternative medical cause. The following age-specific requirements apply:

  * Women < 50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and if they have luteinizing hormone and follicle-stimulating hormone levels in the post-menopausal range for the institution or underwent surgical sterilization (bilateral oophorectomy or hysterectomy).
  * Women ≥ 50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of all exogenous hormonal treatments, had radiation-induced menopause with last menses >1 year ago, had chemotherapy-induced menopause with last menses >1 year ago, or underwent surgical sterilization (bilateral oophorectomy, bilateral salpingectomy or hysterectomy).
* Highly effective contraception for both male subjects and female subjects of child bearing potential throughout the study and for at least 4 months after last study treatment administration (see Section 7.6).
* Recovery to baseline or ≤ Grade 1 CTCAE v5.0 from toxicities related to any prior treatments, unless AE(s) are clinically non-significant and/or stable on supportive therapy.
* Able to provide informed consent and willing to sign an approved consent form that conforms to federal and institutional guidelines.

Exclusion Criteria:

* Subject has received systemic antineoplastic therapy (including unconjugated therapeutic antibodies and toxin immunoconjugates) or any investigational therapy ≤ 14 days or within 5 half-lives prior to starting study treatment, whichever is shorter.
* Subject has received radiotherapy ≤ 14 days prior to the first dose of study treatment. Localized radiation therapy for the treatment of symptomatic bone metastasis is allowed during that timeframe.
* Subjects who have undergone major surgery ≤ 3 weeks prior to starting study drug or who have not fully recovered from major surgery.
* Presence of peritoneal carcinomatosis (PC).
* Diagnosis of any other malignancy within 2 years prior to study enrollment, except for adequately treated basal cell or squamous cell skin cancer, carcinoma in situ of the breast, bladder or of the cervix, and low-grade (Gleason 6 or below) prostate cancer on surveillance with no plans for treatment intervention (eg, surgery, radiation, or castration) or prostate cancer that has been adequately treated with prostatectomy or radiotherapy and currently with no evidence of disease or symptoms is allowed.
* Known brain metastases or cranial epidural disease.

  --Note: Brain metastases or cranial epidural disease adequately treated with radiotherapy and/or surgery and stable for at least 4 weeks before the first dose of study treatment will be allowed on trial. Subjects must be neurologically asymptomatic and without corticosteroid treatment at the time of first dose of study treatment.
* History or current evidence of retinal vein occlusion (RVO) or current risk factors for RVO (e.g. uncontrolled glaucoma or ocular hypertension, history of hyperviscosity or hypercoagulability syndromes).
* Current evidence of uncontrolled, significant intercurrent illness including, but not limited to, the following conditions:

  * Cardiovascular disorders:
  * Congestive heart failure New York Heart Association Class 3 or 4, unstable angina pectoris, serious cardiac arrhythmias.
  * Stroke (including transient ischemic attack [TIA]), myocardial infarction (MI), or other ischemic events, or thromboembolic event (eg, deep venous thrombosis, pulmonary embolism) within 3 months before first dose.
  * QTc prolongation defined as a QTcF > 500 ms.
  * History of seizures
  * Impairment of gastrointestinal function or gastrointestinal disease (e.g., ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection under the judgment of the PI may impair absorption of study drugs).
  * Any other condition that would, in the Investigator's judgment, contraindicate the patient's participation in the clinical study due to safety concerns or compliance with clinical study procedures, e.g., infection/inflammation, intestinal obstruction, unable to swallow medication.(patients may not receive drug through a feeding tube), social/ psychological issues, etc.
* Known HIV infection with a detectable viral load within 6 months of the anticipated start of treatment.

  --Note: Patients on effective antiretroviral therapy with an undetectable viral load within 6 months of the anticipated start of treatment are eligible for this trial.
* Active infection including tuberculosis (clinical evaluation that includes clinical history, physical examination, radiographic findings, and TB testing in line with local practice), hepatitis B (known positive HBV surface antigen (HBsAg) result), or hepatitis C.

  --Note: Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. Patients positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA.
* Medical, psychiatric, cognitive or other conditions that may compromise the patient's ability to understand the patient information, give informed consent, comply with the study protocol or complete the study.
* Known prior severe hypersensitivity to investigational product or any component in its formulations (NCI CTCAE v5.0 Grade ≥ 3).
* Subjects taking prohibited medications as described in Section 6.4. A washout period of prohibited medications for a period of at least 5 half-lives or as clinically indicated should occur prior to the start of treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2020-03-17 (Actual); Primary Completion 2022-06-10 (Actual); Study Completion 2022-08-18 (Actual)

PRIMARY OUTCOMES:
Recommended phase 2 dose of ulixertinib in combination with a fixed dose of hydroxychloroquine in subjects with advanced, RAS, non-V600 BRAF, ERK or MEK mutated gastrointestinal malignancies | the day of the first dose, cycle one day one, to cycle one day 28 (Cycle=28 days)
  The incidence of DLTs during the defined DLT period

SECONDARY OUTCOMES:
Safety and tolerability of ulixertinib and hydroxychloroquine in the study population: adverse events (AEs) and serious adverse events (SAEs) | Any patient who has taken at least one dose of both ulixertinib and hydroxychloroquine will be evaluable for toxicity. Assessment will be completed through safety follow-up visit at 60 days after the end of treatment visit.
  The frequency of adverse events (AEs) and serious adverse events (SAEs) characterized by type, severity (as defined by the NIH CTCAE, version 5.0), seriousness, duration, and relationship to study treatment
Efficacy of ulixertinib and hydroxychloroquine in the study population: Objective response rate (PR and CR) | Patients will be evaluable for response once they have completed the first cycle of treatment and completed the C2D1 CT Scan.Assessment will be completed through safety follow-up visit at 60 days after the end of treatment visit.
  Objective response rate (PR and CR) will be described

CONTACTS AND LOCATIONS:
Locations (1):
- Huntsman Cancer Institute, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No